CLINICAL TRIAL: NCT01359826
Title: The Effect of Milnacipran on Fatigue and Quality of Life in a Lupus Cohort
Brief Title: The Effect of Milnacipran on Fatigue and Quality of Life in Lupus Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI has let the institution. We are unable to locate any study documents that would indicate study enrollment
Sponsor: Loma Linda University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5110068
Record Dates: First submitted 2011-04-19; First posted 2011-05-25 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Systemic Lupus Erythematosus; Widespread Pain; Fibromyalgia
Keywords: Systemic Lupus Erythematosus; Widespread Pain; Fibromyalgia; Fatigue; Pain; Quality of Life
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Fibromyalgia; Fatigue; Pain | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Milnacipran (Experimental): Patients administered milnacipran will receive a dose escalation to 50 mg twice a day over 12 days and continued at this dose until week 6. If tolerated and a 15% improvement in fatigue from baseline is achieved by assessment on the FSS, then patients will continue taking 50 mg twice a day until the end of the study on day 98 (week 14). Otherwise, the dose of milnacipran will be titrated upward to 100 mg twice a day over 12 days and continued at this dose until day 98 (week 14).
  Interventions: Drug: Milnacipran
- Placebo (Placebo Comparator): Placebo tablets administered orally twice a day for 14 weeks.
  Interventions: Drug: Milnacipran

INTERVENTIONS:
Drug: Milnacipran — After dose escalations, patients will receive Milnacipran administered at 50 mg twice a day after for 12 weeks or milnacipran 50 mg twice day for 4 weeks and then 100 mg twice a day for an additional 6 weeks depending on tolerability and fatigue response.
  Other Names: Savella

SUMMARY:
Systemic lupus erythematosus (SLE) is a chronic multi-system autoimmune disease impacting the physical, social, psychological health and quality of life of patients. Fatigue and pain are aspects of SLE patients which affect their health related quality of life (HRQOL). The purpose of this study is to determine the effect of milnacipran on fatigue in SLE patients with widespread pain (WSP) or fibromyalgia syndrome (FMS). A secondary objective will be to determine the effect of milnacipran on pain and quality of life measurements. Fifty SLE male and female patients, 18 years and older, will be recruited for a 15-week study, in which patients will be receive 14 weeks of milnacipran 50-100 mg twice a day or placebo. Measurements of fatigue, pain, and HRQOL will be compared between the milnacipran and placebo groups at the screening visit, baseline visit, week number 6, and week number 14. Milnacipran has been shown to be an effective treatment for pain, fatigue and physical function in FMS patients. To date, no clinical trials have demonstrated efficacy for the treatment of fatigue in SLE patients with concomitant WSP or FMS. The investigators hypothesize, based on FMS studies, that the milnacipran treated patients will have less fatigue than those in the placebo group. In addition, compared to control arm, those treated with the study drug will have less pain and improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Female or male age 18 or older.
* Has fulfilled the 1997 classification criteria for SLE.
* Has chronic WSP or FMS.
* Score a 40 or more on the visual analog score (VAS) for fatigue.

Exclusion Criteria:

* Has a chronic inflammatory autoimmune condition other than SLE.
* Has an acute or uncontrolled co-morbid medical condition.
* Uncontrolled narrow angle glaucoma.
* Has been hospitalized in the last four months for a lupus flare.
* Pregnant or breast feeding.
* Has a current or prior major depressive disorder or other DSM IV diagnosis within 2 years of the screening visit.
* The use of antidepressants, MAO inhibitors, antipsychotics or lithium
* The use of pregabalin or milnacipran within 2-4 weeks.
* Has received cyclophosphamide and or rituximab within 4 and 6 months.
* Unable to speak, read, and understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Fatigue | Baseline and Week 14
  A change in fatigue from baseline will be assessed with values obtained at week 14 using the Fatigue Severity Scale (FSS) in both the treatment and control groups.

SECONDARY OUTCOMES:
Fatigue | Baseline and Week 6
  A change in fatigue will be assessed with values obtained at baseline and week 6 using the FSS and Visual Analogue Score (VAS) Fatigue.
Pain | Baseline, week 6 and week 14
  A change in pain will be assessed with values obtained at baseline, week 6, and 14 using the VAS Pain, and the Short Form - McGill Pain Questionnaire (SF-MPQ).
Health related quality of life | Baseline, week 6 and week 14
  Health related quality of life will be assessed with values obtained at baseline, week 6, and 14 using the Short form-36 (SF-36).
Overall health status | Baseline, week 6 and week 14
  A change in overall health status will be assessed using the Patient Global Impression of Change (PGIC) at baseline, week 6, and 14.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel P. Katsaros, D.O., Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States